CLINICAL TRIAL: NCT06625190
Title: Allogeneic Stem Cell Transplantation Utilizing Alpha/Beta T Cell and CD19+ B Cell Depletion With Zoledronic Acid in Combination to Treat Pediatric, Adolescent, and Young Adult Patients With Relapsed/Refractory Solid Tumors
Brief Title: Alpha/Beta T and B Cell Depletion With Zoledronic Acid for Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: UF-PED-006; IRB202500132 (Other: University of Florida)
Record Dates: First submitted 2024-10-01; First posted 2024-10-03 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Neuroblastoma; Rhabdomyosarcoma; Synovial Sarcoma; Peripheral Nerve Sheath Tumors; Clear Cell Sarcoma; Alveolar Soft Part Sarcoma; Desmoplastic Small Round Cell Tumor; Chordoma; Rhabdoid Tumor; Epithelioid Sarcoma; Myoepithelial Tumor; Osteosarcoma; Ewing Sarcoma
Keywords: pediatric solid tumors; stem cell transplantation; graft manipulation
MeSH Terms: conditions — Neuroblastoma; Rhabdomyosarcoma; Sarcoma, Synovial; Nerve Sheath Neoplasms; Sarcoma, Clear Cell; Sarcoma, Alveolar Soft Part; Desmoplastic Small Round Cell Tumor; Chordoma; Rhabdoid Tumor; Sarcoma; Myoepithelioma; Osteosarcoma; Sarcoma, Ewing | interventions — Zoledronic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- alpha/beta T cell and CD19+ B cell depleted stem cell graft with zoledronic acid (Experimental)
  Interventions: Device: Miltenyi CliniMACS Prodigy ® system; Drug: Zoledronic acid

INTERVENTIONS:
Device: Miltenyi CliniMACS Prodigy ® system — Subjects will receive an allogeneic stem cell transplant that has been depleted of ⍺/β T-cells and CD19+ B-cells using the Miltenyi CliniMACS Prodigy® system.
Drug: Zoledronic acid — All subjects will receive zoledronic acid intravenously on days +28, +56, +84, +112, and +140.
  Dosing in the phase Ib portion of the study will follow a 3 + 3 design where the first 3 subjects will receive the expected phase II dose of 1.25 mg/m2 (dose level 1). If no dose-limiting toxicities (DLTs) occur in these subjects, dose level 1 will be the maximum tolerated dose. However, if at least 1 DLT is observed in the first 3 patients, 3 additional subjects will be enrolled at dose level 1. If more than 2 DLTs are observed in these 6 subjects, then dose de-escalation to 0.8 mg/m2 (dose level 0) will occur and 3-6 additional subjects may be enrolled.
  All subjects in the phase II portion of the study will receive the maximum tolerated dose determined in the phase Ib portion.

SUMMARY:
Hematopoietic stem cell transplantation can cure patients with blood cancer and other underlying diseases. αβ-T cell and B cell depletion has been introduced to decrease GVHD and PTLD and has demonstrated effectiveness for hematologic malignancies and non-malignant diseases additionally increasing the donor pool as to allow for haploidentical transplant to safely occur.

While solid tumors can be highly chemotherapy sensitive, many remain resistant and require multimodalities of treatment. Immunotherapy has been developed to harness the immune system in fighting solid tumors, though not all have targeted effects. Some solid tumors are treated with autologous transplants; however, they do not always demonstrate an improved event free survival or overall survival. There has been evidence of the use of allogeneic stem cell transplants to provide a graft versus tumor effect, though studies remain limited.

By utilizing αβ-T cell and B cell depletion for stem cell transplants and combining with zoledronic acid, the immune system may potentially be harnessed and enhanced to provide an improved graft versus tumor effect in relapsed/refractory solid tumors and promote an improved event-free survival and overall survival.

This study will investigate the safety of treatment with a stem cell graft depleted of αβ-T cell and CD19+ B cells in combination with zoledronic acid in pediatric and young adult patients with select solid tumors, as well as whether this treatment improves survival rates in these patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients 6 months to ≤ 25 years old
* Relapsed/Refractory Solid Tumor whom failed or deemed ineligible to receive autologous transplant or if autologous transplant did not offer >20% chance of cure with the following diseases:

  1. neuroblastoma (high risk with relapsed or refractory disease),
  2. relapsed/refractory rhabdomyosarcoma,
  3. relapsed/refractory non-rhabdomyosarcoma soft tissue sarcoma (NRSTS): synovial sarcoma, malignant peripheral nerve sheath tumors (MPNST),
  4. High risk adult type NRSTS: clear cell sarcoma, alveolar soft part sarcoma,
  5. Other high-risk extracranial solid tumors: desmoplastic small round cell tumors, chordoma, malignant rhabdoid tumor, epithelioid sarcoma, myoepithelial tumor
  6. relapsed/refractory bone tumors: osteosarcoma and Ewing sarcoma/PNET, or
  7. other high-risk solid tumors with <10% expected survival with conventional treatment.
* Subjects must not have more than one active malignancy at the time of enrollment. (Subjects with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen [as determined by the treating physician and approved by the PI] may be included.)
* Haplo-identical related donor (at least one full haplotype must be matched).
* Karnofsky or Lansky score ≥60% at the time of enrollment. Karnofsky scores must be used for patients >16 years of age and Lansky scores for patients ≤16 years of age
* Adequate organ function (within 4 weeks of initiation of preparative regimen), defined as:

  1. Pulmonary: FEV1, FVC, and corrected DLCO must all be ≥ 50% of predicted by pulmonary function tests (PFTs). For children who are unable to perform for PFTs due to age, the criteria are: no evidence of dyspnea at rest and no need for supplemental oxygen.
  2. Renal: Creatinine clearance or radioisotope GFR ≥60 mL/min/1.73 m2 or a serum creatinine based on age/gender
  3. Cardiac: Ejection fraction of ≥ 40% by echocardiogram or radionuclide scan (MUGA).
* Written informed consent obtained from the subject and the subject agrees to comply with all the study-related procedures
* Individuals of childbearing potential (IOCBP) must be using an adequate method of contraception to avoid pregnancy throughout the study and for one year following transplantation to minimize the risk of pregnancy. Prior to study enrollment, individuals of childbearing potential must be advised of the importance of avoiding pregnancy during trial participation and the potential risk factor for an unintentional pregnancy.
* Subjects with female partners of child-bearing potential must agree to use physician-approved contraceptive methods (e.g., abstinence, condoms, vasectomy) throughout the study and should avoid conceiving children for one year following stem cell transplantation.

Exclusion Criteria:

* Patients with documented uncontrolled infection at the time of study entry are not eligible.

  a. Uncontrolled infection is patient without treatment antimicrobials and/or demonstrating progression despite antimicrobials
* Demonstrated lack of compliance with medical care, as determined by the treating physician.
* Patients who have received an allogeneic HSCT within 6 months.
* Patients who do not have an eligible allogeneic donor available.
* Patients with a life expectancy <3 months
* Patients not meeting inclusion criteria for organ function.
* Females or males of childbearing potential who are unwilling or unable to use an acceptable method to avoid pregnancy for the entire study period and for at least one year after transplantation.
* Females who are known to be pregnant or breastfeeding.
* History of any other disease, metabolic dysfunction, clinical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of protocol therapy or that might affect the interpretation of the results of the study or that puts the subject at high risk for treatment complications, in the opinion of the treating physician.
* Prisoners or subjects who are involuntarily incarcerated, or subjects who are compulsorily detained for treatment of either a psychiatric or physical illness.

Ages: 6 Months to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 27 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2030-02 (Estimated); Study Completion 2030-02 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival rate | 1 year post-transplant
  Determine the disease-free survival rate at 1 year post-transplant
Incidence of aGVHD | 2 years post-transplant
  Determine the incidence of grade II-IV acute graft versus host disease (aGVHD)

SECONDARY OUTCOMES:
Disease-free survival rate | 100 days post-transplant
  Determine the disease-free survival rate at 100 days post-transplant
Disease-free survival rate | 2 years post-transplant
  Determine the disease-free survival rate at 2 years post-transplant
Overall survival rate | 100 days post-transplant
  Determine the overall survival rate at 100 days post-transplant
Overall survival rate | 1 year post-transplant
  Determine the overall survival rate at 1 year post-transplant
Overall survival rate | 2 years post-transplant
  Determine the overall survival rate at 2 years post-transplant

CONTACTS AND LOCATIONS:
Overall Officials: Jordan Milner, MD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States